CLINICAL TRIAL: NCT02057081
Title: Multifamily Group to Reduce Marital Conflict and Disability in Veterans With mTBI
Acronym: MFG-mTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1106-R; 1I01RX001106 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-02-06 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Mild Traumatic Brain Injury; Posttraumatic Stress Disorders; Depression
Keywords: Stress Disorders, Post-traumatic; Mild Traumatic Brain Injury; Veterans Health; Veterans; Spouses; Couples; Psychotherapy, Group; Depression; Couples Therapy; Family Therapy; PTSD; posttraumatic stress disorder
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic; Depression | interventions — Family Characteristics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Intensive 14-session psychoeducational rehabilitation and skills-building intervention for couples.
  Interventions: Behavioral: Multifamily Group for mTBI for Couples
- Control (Active Comparator): Didactic 14-session educational group intervention for families.
  Interventions: Behavioral: Group Health Education (GHE)

INTERVENTIONS:
Behavioral: Multifamily Group for mTBI for Couples — MFG-mTBI-C uses a structured problem-solving and skills training approach to provide Veterans and partners with tools and information to improve coping and help couples reconnect through positive behavioral exchanges.
  Other Names: MFG-mTBI-C
  Arms: Treatment
Behavioral: Group Health Education (GHE) — GHE is a 14-session, highly structured educational intervention providing general information on health problems that are common among the general OEF/OIF cohort including sleep and sleep problems, physical activity and exercise, and alcohol and drug use, as well as guidelines for improving health behavior in these areas.
  Other Names: GHE
  Arms: Control

SUMMARY:
This project addresses the rehabilitation and mental health needs of married combat Veterans post-deployed from Iraq or Afghanistan with a mild traumatic brain injury (mTBI) and/or significant posttraumatic stress (PTS) or combat-related stress (CS) by providing psychoeducation, communication and problem solving skills in a multifamily group (MFG) setting. In this group, Veterans and spouses/cohabiting partners learn customized therapeutic strategies to help compensate for deficits and promote Veteran community integration, interpersonal and emotion regulation skills, and marital satisfaction. The effectiveness of the skills-based MFG will be compared to that of a health education group which offers a supportive environment and basic education without skills training through a randomized clinical trial. As there is currently no family-based intervention for Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans with mTBI offered within the VA spectrum of services, this intervention fills a crucial gap in healthcare for our newest Veterans.

DETAILED DESCRIPTION:
Mild traumatic brain injury (mTBI), an injury or concussion associated with brief loss of consciousness or altered mental state, has affected as many as 35% of soldiers wounded during recent military actions in Iraq and Afghanistan. Up to 30% of those injured report persistent somatic, emotional and cognitive post-concussive symptoms (PCS) which may adversely impact family life and community re-integration. Marital conflict and intimate partner violence, reported by 54% of OEF/OIF couples, and co-occurring mental health problems may exacerbate cognitive dysfunction and delay rehabilitation. A key contributor to marital conflict is a lack of knowledge about the Veteran's condition and the skills needed to help him compensate for common deficits in memory and planning which create challenges in household management. Despite a growing evidence base for couples treatment for PTSD, there is no established family-based treatment for OEF/OIF Veterans with mTBI, creating a critical research and services gap. The proposed research aims to fill this gap by evaluating a novel form of multi-family group treatment designed to improve community integration (CI) among married/cohabiting OEF/OIF Veterans with mTBI and/or significant posttraumatic stress (PTS) or combat-related stress (CS) by training spouse/partners to aid with rehabilitation and employing disability-adapted communication and problem-solving skills to reduce marital conflict and improve marital satisfaction.

Veterans (N=150) with a positive Defense and Veterans Brain Injury Center (DVBIC) screen for mTBI sustained during the OEF/OIF era, confirmed by the VA Identification Clinical Interview and a Montreal Cognitive Assessment (MoCA) score 19 or if they either meet diagnostic criteria for PTSD or have trauma- or CS of at least moderate severity, as defined by either a) PTSD Checklist (PCL) score >34 or b) Customer Effort Score (CES) score of >23, will be randomized to receive either: 1) Multifamily Group for TBI for Couples (MFG-mTBI-C), a psychoeducational, rehabilitation and skills-building intervention consisting of a 2-session multifamily educational workshop providing information about TBI and 12 bi-monthly multifamily group meetings providing skills training in problem-solving and communication related to cognitive/emotional deficits; or 2) 14 bi-monthly multifamily group sessions delivering health education without skills training. Both treatments will be preceded by 2-3 individual couples sessions. Participants will be assessed pre- and post-treatment and 6 months post-treatment. Data will be analyzed using an intent-to-treat analysis with paired comparisons between treatment groups on primary (Veteran CI, caregiver burden) and secondary (anger management, use of social supports) outcome variables using mixed effects regression models. It is hypothesized that Veterans treated with MFG-mTBI-C will show improved CI, anger management and use of social support, and spouse/partners will show reduced burden compared with those treated in the health education group. If efficacious, MFG-mTBI-C has the potential to assist Veterans with mTBI and their partners throughout the VA Health Care System.

ELIGIBILITY:
Inclusion Criteria:

Eligible Veterans must have a diagnosis of mTBI in accordance with the VA/DoD Clinical Practice Guideline for Management of Concussion/Mild Traumatic Brain Injury: injury or concussion associated with at least one of the following: brief (< 30 minutes) loss of consciousness or altered state of consciousness or post-traumatic amnesia for < 24 hours following the injury, or they either meet diagnostic criteria for PTSD based on the MINI or have trauma- or CS of at least moderate severity, as defined by either: a) PCL score >34; or b) CES score of >23.

* The TBI must be either blast-related or attributable to another discrete event (e.g., fall, fight, injury) sustained during deployment in the OEF/OIF era.
* Post-concussive symptoms (e.g., sleep or memory problems, headache) must not be attributable to a subsequent injury or other pre-existing or concurrent neurologic disorder:
* Eligible Veterans must also have a consenting, qualifying spouse/cohabiting partner and a Montreal Cognitive Assessment (MoCA) (Nasreddine,2005) score 19.
* The 30-item MoCA screens for impairment in specific areas of cognitive functioning deemed necessary for participation in a 90-minute, structured group including attention and concentration, executive functions, language and conceptual thinking.
* We have specified a MoCA cut-off at the lower end of the range for mild cognitive dysfunction (19), in order to exclude Veterans with severe memory and/or other cognitive deficits, while admitting those with more mild deficits, as these represent our target population, i.e. Veterans with a history of mTBI.

Inclusion criteria-partners: Legally married to or co-residing with Veteran for at least 6 months, with no plans for divorce or separation.

Exclusion Criteria:

Exclusion criteria for Veterans and partners are:

* a lifetime diagnosis of a major psychiatric disorder (schizophrenia, schizoaffective or bipolar disorder with psychotic features) or active psychosis based on the Structured Clinical Interview for DSM-IV-TR (SCID-L) (First et al., 2007).
* alcohol or drug abuse or dependence with past 6 months defined by a Short Michigan Alcoholism Screening Test (SMAST) (Selzer, 1975) 3, based on the recommended cut-off for TBI survivors (Gentilello et al.,1995) or a Drug Abuse Screening Test-10 (DAST-10) (Skinner, 1982) 3.
* "severe" inter-partner violence as defined by the revised 20-item Conflict Tactics Scale Short Form (CTS2S) (Straus & Douglas, 2004).
* a suicide attempt within the past 6 months (aborted and interrupted attempts) as assessed by the Columbia Suicide Severity Rating scale (C-SSRS).
* medical condition or life event (e.g., ongoing or pending legal action in another state) that would compromise participation.
* participation of either the caregiver or Veteran in another psychosocial intervention trial or couples' treatment six months prior to or during study or follow-up. Participation in individual psychotherapy and pharmacotherapy are permitted: use of and starting/stopping these services will be tracked. Participants will be screened for inclusion/exclusion as described above immediately after giving consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Drapalski, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (3):
- United States (3):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was consented but their partner did not consent.
Period: Overall Study
Arm/Group | Treatment | Control
Started (Includes both veteran and partner participants) | 136 | 112
Completed Baseline (Veterans and partners who were consented, randomized, completed baseline and deemed eligible) | 88 | 80
Post-Treatment Assessment (Includes both veteran and partner participants) | 58 | 52
Completed (Includes both veteran and partner participants) | 46 | 44
Not Completed | 90 | 68

BASELINE CHARACTERISTICS:
Population: Reflects demographic characteristics of those participants who consent, were randomized and completed the baseline assessment (does not include those that were enrolled and did not complete or who were ineligible)
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 88 | 80 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age is missing for one participant assigned to the experimental treatment condition
  years
    number analyzed (Participants) | 87 | 80 | 167
    (all) | 37.7 (9.1) | 36.2 (9.2) | 37.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 84
  Male | 44 | 40 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 32 | 24 | 56
  White | 44 | 36 | 80
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 3 | 12 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88 | 80 | 168
Relationship Status [Count of Participants; unit: Participants]
  Married | 56 | 50 | 106
  Cohabitating | 24 | 24 | 48
  Engaged | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in the Community Reintegration of Injured Service Members Computer Adaptive Test (CRIS-CAT)
Description: The Community Reintegration of Injured Service Members Computer Adaptive Test (CRIS-CAT) was used to measure community reintegration. The measure includes 3 subscales: Extent of Participation, Perceived Limitations, and Satisfaction. A total score for each subscale is calculated by summing item responses (range= 10 to 140), with higher scores indicating greater frequency of community participation (extent of participation), greater perceived limitations to community participation (perceived limitations), and greater satisfaction with community participation (satisfaction).
Time Frame: baseline, post-treatment in study month 38 after 12 bimonthly sessions, and 6-months post-treatment in study month 44
Population: Only veteran participants were administered and evaluated on this outcome (not their partners). Two participants from the treatment group and 3 participants from the control group were missing data for this outcome at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 42 | 37
score on a scale
  Baseline: Extent of Participation Subscale | 36.4 (7.8) | 35.0 (5.4)
  Post-Treatment: Extent of Participation Subscale: number analyzed (Participants) | 24 | 19
  Post-Treatment: Extent of Participation Subscale | 38.2 (6.4) | 35.1 (6.1)
  6-Month Follow-Up: Extent of Participation Subscal: number analyzed (Participants) | 20 | 16
  6-Month Follow-Up: Extent of Participation Subscal | 37.6 (7.9) | 38.0 (6.5)
  Baseline: Perceived Limitations Subscale: number analyzed (Participants) | 41 | 36
  Baseline: Perceived Limitations Subscale | 41.0 (4.9) | 41.0 (4.9)
  Post-Treatment: Perceived Limitations Subscale: number analyzed (Participants) | 24 | 19
  Post-Treatment: Perceived Limitations Subscale | 41.7 (5.1) | 41.3 (4.8)
  6-Month Follow-Up: Perceived Limitations Subscale: number analyzed (Participants) | 20 | 16
  6-Month Follow-Up: Perceived Limitations Subscale | 41.1 (4.7) | 42.3 (4.5)
  Baseline: Satisfaction Subscale: number analyzed (Participants) | 41 | 36
  Baseline: Satisfaction Subscale | 39.8 (6.0) | 39.9 (4.5)
  Post-Treatment: Satisfaction Subscale: number analyzed (Participants) | 24 | 19
  Post-Treatment: Satisfaction Subscale | 41.0 (5.7) | 40.3 (4.7)
  6-Month Follow-Up: Satisfaction Subscale: number analyzed (Participants) | 20 | 16
  6-Month Follow-Up: Satisfaction Subscale | 39.3 (3.4) | 38.9 (7.9)

2. Secondary Outcome: Change in Caregiver Burden Inventory
Description: The Caregiver Burden Inventory is a 24-item scale that measures caregiver burden in four areas: physical, social, emotional and time dependence burden. A total score is calculated by summing the item responses (range= 1 to 100), with higher scores indicating greater caregiver burden.
Time Frame: Baseline, post-treatment in study month 38 after 12 bimonthly sessions, and 6-months post-treatment in study month 44
Population: Only partner/spouse participants were administered and evaluated on this outcome (not veterans).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 44 | 40
score on a scale
  Baseline | 24.9 (20.0) | 25.8 (16.5)
  Post-treatment: number analyzed (Participants) | 26 | 23
  Post-treatment | 24.8 (22.3) | 25.6 (15.0)
  6-month Post-Treatment: number analyzed (Participants) | 19 | 20
  6-month Post-Treatment | 21.5 (19.0) | 27.1 (20.1)

ADVERSE EVENTS:
Time Frame: Duration of participants involvement in the study, up to ~ 16 months
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/112
Serious Adverse Events (participants affected / at risk) | 6/136 | 4/112
Other Adverse Events (participants affected / at risk) | 0/136 | 0/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=136) | Control (N=112)
self-reported interpersonal violence (Social circumstances) | 3 | 0 — Self-reported physical altercation with partner
psychiatric hospitalization (Psychiatric disorders) | 0 | 1
medical hospitalization (Surgical and medical procedures) | 1 | 0
Medical hospitalization (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Medical hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Medical hospitalization (Immune system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT02057081/Prot_SAP_000.pdf